CLINICAL TRIAL: NCT04714723
Title: Lifestyle Intervention Trial in High Metabolic Risk Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAS-LIT-202101
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: weight loss,metabolic risk, lifestyle intervention, homeostasis
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmed smartphone intervention group (Active Comparator): Subjects will receive programmed-smartphone lifestyle intervention
  Interventions: Behavioral: Programmed smartphone intervention
- Programmed smartphone plus dietitian intervention group (Experimental): Subjects will receive programmed-smartphone plus dietitian lifestyle intervention
  Interventions: Behavioral: Programmed smartphone plus dietitian intervention

INTERVENTIONS:
Behavioral: Programmed smartphone intervention — Interactive programmed lifestyle education based on smartphone for six month
  Arms: Programmed smartphone intervention group
Behavioral: Programmed smartphone plus dietitian intervention — Interactive programmed lifestyle education based on smartphone plus dietitians support for six month
  Arms: Programmed smartphone plus dietitian intervention group

SUMMARY:
In this single-blind, randomized trial, 395 eligible volunteers, who have higher metabolic syndrome (MetS) risk and aged 20-65 years, will be assigned to one of two smartphone-based lifestyle intervention arms: 1) Programmed-smartphone intervention or 2) Programmed-smartphone plus dietitian intervention. Before and after 6-month intervention, "PhenFlex test" (PFT) was performed to examine and quantify improved metabolic flexibility.

This intervention trial will be conducted by researchers in Shanghai Institute of Nutrition and Health of the Chinese Academy of Sciences (CAS) collaborating with Zhejiang University affiliated Sir Run Run Shaw Hospital. The study protocol was approved by the Ethics Committees in Shanghai Institutes of Nutrition and Health, and in Sir Run Run Shaw Hospital.

The main aims of this study are to determine 1) efficacy of lifestyle interventions with different intensity in reducing MetS and its risk factors; 2) improved metabolic responses or flexibility defined by PFT-based homeostasis index; and 3) major genetic and nongenetic determinants for the efficacy of interventions among high MetS risk Chinese.

DETAILED DESCRIPTION:
Metabolic syndrome, a cluster of multiple metabolic disturbances, including central obesity, dyslipidemia, hypertension, and hyperglycemia, is associated with 2-5-fold heightened risks of CVD and T2D. Compelling evidence showed that lifestyle intervention is one of effective approaches for preventing and controlling cardiometabolic diseases. However, there were considerably variations among different interventions and different persons. With widely available smartphone and APP-connected wearable devises, it is possible to provide programmed nutrition and lifestyle education to help participants achieve intervention targets, and closely monitor compliance. However, few studies investigated the efficacy of lifestyle interventions with programmed smartphone and APP-connected wearable devises in MetS management. Moreover, since present disease-based diagnoses and biomarkers may not adequately define health status, the concept of "re-redefining health" has attracted growing attention. The phenotypic flexibility and "PhenFlex test" are one of approaches to measure individuals' adaptive capacity to maintain hemostatic condition after having a standardized challenge drinker. To date, the PFT has been studied among 10,000 subjects in western countries and few studies, if any, have conducted in Chinese who have different genetic background and dietary patterns. It remains to be established whether and to what extent that the PFT-based hemostatic index system can precisely evaluate the metabolic health in Chinese.

In the current trial, 395 subjects with MetS risks were randomly assigned to either smartphone-based lifestyle intervention arms: 1) Programmed-smartphone intervention; or 2) Programmed-smartphone plus dietitian intervention. The intervention duration will be 6-month and then have 2-year follow-up. During starting and end of 6-month intervention, we included PFT during the physical examination hold in the Sir Run Run Shaw Hospital. All the subjects were given a standardized challenge drinker (75g glucose, 60 fat and 20g protein). Fasting and multiple postprandial time points samples (blood, t=0,1,3h) and urine and feces were collected to measure clinical and omics markers like metabolomics, gut microbiota and SNPs. Finally, the homeostasis index will be built to estimate improvement of individual metabolic health after the intervention. In conclusion, this study will provide scientific evidence and novel insights about the effectiveness of new intervention strategies and precise diagnostic and assessment system for cardiometabolic management.

ELIGIBILITY:
Inclusion Criteria:

Volunteers at high metabolic risk aged 20-65 who didn't participate in other studies in 3 months before the current research, having a certain level of education and normal cognitive ability, taking good care of himself/herself. MetS risk factors were identified by the definition proposed by the International Diabetes Federation criteria for Chinese adults. Participants should have central obesity (waist circumference ≥90 cm in men or ≥80 cm in women).

Exclusion Criteria:

* Fasting glucose>7.0mmol/L after taking insulin or other blood glucose-lowering drugs
* Diagnosed phase three hypertension or can't lowering SBP under 160mmHg after anti-hypertension drugs
* Fasting blood TG≥ 5.7 mmol/L or fasting LDL-C≥ 4.9 mmol/L after taking lipid-lowering drugs
* Pregnancy or lactation
* Obvious drug changing in three months before research
* History of drug or alcohol abuse or other substance abuse (Alcohol abuse is defined as more than 40 g/day of alcohol for woman, and more than 80g/day for man)
* Severe kidney and liver diseases (blood biomarkers such as alt, serum creatinine is 1.5 times over the scope of normal setting)
* Severe Gastrointestinal diseases (such as severe diarrhea, constipation, severe digestive tract inflammation, active peptic ulcer, acute cholecystitis, etc.)
* Having surgeries within one year before research such as heart stents implanted surgery (expect for appendicitis or hernia operation)
* Severe cardiovascular disease (e.g., heart failure, myocardial infarction, cerebral infarction, and acute myocarditis, severe arrhythmia, received the intervention therapy, etc.)
* Cancer or receiving radiotherapy and chemotherapy within 5 years
* Severe pituitary or thyroid diseases
* Suffering from AIDS, hepatitis A, hepatitis B and other infectious diseases
* Mental disorders or current use of antidepressants

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline and month 6
  Weight will be assessed by Seca-255 (ScalesGalore) during each visit ,weight will also be assessed by Bluetooth scale at home

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline and month 6
  Body mass index (BMI) will be assessed by Seca-201(ScalesGalore) during each visit
Waist circumference | Baseline and month 6
  Waist circumference will be assessed by Seca-201(ScalesGalore) during each visit
Blood pressure | Baseline and month 6
  Both systolic pressure and diastolic pressure will be assessed using electronic blood pressure monitor (Omron J750)during each visit and at home
Triglyceride | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Total cholesterol | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
LDL-C | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
HDL-C | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Glucose | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Metabolic Homeostasis Score | Baseline and month 6
  A metabolic homeostasis score is a composite score that includes aggregated changes in blood biomarkers (metabolites or biomarkers or index involved in carbohydrates metabolism such as glucose, C-peptide, Matsuda index etc.; metabolites or biomarkers involved in lipid metabolism such as high-density lipoprotein cholesterol, total cholesterol, triglyceride etc.; metabolites or biomarkers involved in protein/vitamin metabolism such as creatinine; inflammatory or cytokines such as interleukin-6 etc.; hormones; anthropometric measures etc.).
  The metabolic homeostasis score is a composite score, that is calculated by the average of the scores of above-mentioned features using a certain computational algorithm. The larger the metabolic homeostasis score is, the worse the homeostatic resilience of the person, and vice versa.
Body composition | Baseline and month 6
  Body composition will be assessed by InBody-720 multi-frequency bioelectrical impedance device.
Compliance | Whole 6-month intervention
  Behavioral compliance will be assessed by wearable devices and bluetooth devices.

OTHER OUTCOMES:
E-selectin concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
P-selectin concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Vascular cell adhesion molecule-1(VCAM-1) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Intercellular adhesion molecule-1 (ICAM-1) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Amyloid A1(SAA1) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Tumor Necrosis Factor-α (TNF-α) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Interleukin-10(IL-10) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Interleukin-1b(IL-1b) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
C-reactive protein(CRP) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Retinol binding protein(RBP4) concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Adiponectin concentration | Baseline and month 6
  Concentration at fasting and postprandial 60min and 3hours will be measured
Metabolomics including profiling of free fatty acids and other metabolites | Baseline and month 6
  Metabolomics will be measured by LC-MS
Single nucleotide polymorphism (SNPs) | Baseline
  Mutations at specific sites will be detected by gene chip
Gut microbiota 16S rDNA sequencing | Baseline and month 6
  Gut microbiota 16S rDNA will be sequenced
HbA1c | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Insulin | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Glucagon | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Glucagon-like peptide-1 | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Aspartate transaminase | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Gastric inhibitory peptide | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Alanine aminotransferase | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Serum creatinine | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
γ-glutamyl transpeptidase | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Urine creatinine | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Urea nitrogen | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured
Uric acid | Baseline and month 6
  Values at fasting and postprandial 60min and 3hours will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Shanghai Institute of Nutrition and Health, Chinese Acadamy of Sciences
Locations (1):
- Sir Run Run Shaw Hospital;Hangzhou Dianzi University;China Jiliang University; Zhejiang Sci-Tech University, Hangzhou, Zhejiang, China